CLINICAL TRIAL: NCT06192888
Title: Pilot Study of Glofitamab and Lenalidomide in Patients With Relapsed or Refractory Mantle Cell Lymphoma Previously Treated With a BTK Inhibitor
Brief Title: A Study of Glofitamab and Lenalidomide in People With Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-319
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma; MCL
Keywords: Mantle Cell Lymphoma; MCL; Memorial Sloan Kettering Cancer Center; 23-319
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — glofitamab; obinutuzumab; Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Mantle Cell Lymphoma (Experimental): Participants will be diagnosed with relapsed, refractory (R/R) mantle cell lymphoma (MCL) with prior BTK inhibitor (BTKi) failure
  Interventions: Drug: Glofitamab; Drug: Obinutuzumab; Drug: Lenalidomide

INTERVENTIONS:
Drug: Glofitamab — IV Glofitamab
Drug: Obinutuzumab — IV Obinutuzumab
Drug: Lenalidomide — Oral Lenalidomide

SUMMARY:
The purpose of this study is to find out whether the combination of glofitamab and lenalidomide is an effective treatment for relapsed or refractory Mantle Cell Lymphoma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing Informed Consent
* ECOG 0-2
* Histologic diagnosis confirmed as relapsed/refractory mantle cell lymphoma according to WHO guidelines, confirmed by the pathology department at the treating institution
* If the patient previously received CD20 directed therapy, there must be evidence of CD20 expression on neoplastic cells according to instutitional pathology department guidelines. This must be confirmed on a biopsy of Relapsed/Refractory Mantle Cell Lymphoma performed after receipt of the last CD20 directed therapy.
* At minimum 10 unstained slides or tissue block from tumor containing FFPE biospecimen sample from a Relapsed/Refractory Mantle Cell Lymphoma biopsy is required for tumor genomic profiling and MRD testing. If adequate archival tissue is not available, then a repeat biopsy will be required. This requirement can be waived (i.e. if site of disease is inaccessible) after discussion with the MSKCC Principal Investigator
* Tumor genomic profiling from a biopsy sample collected within 6 months of signing informed consent form is required. For MSK patients, this will be done via MSK IRB#12-245 (Integrated Mutation Profiling of Actionable Cancer Targets (IMPACT)) within 6 months prior to signing Informed Consent form, and preferably repeated for patients who did not have IMPACT performed after discontinuing their last line of treatment. Patients at external sites will run genomic profiling per institutional guidelines. If sites do not have an approved assay available, they may send archival tissue to MSK. Details included in lab manual
* Previously treated with at least one prior line of systemic therapy for mantle cell lymphoma. Prior BTKi failure is required. BTKi failure is defined as progression of disease during BTKi therapy or patients must have progressed or relapsed after completing BTK inhibitor therapy, or failed to achieve a PR following 12 weeks of BTK inhibitor therapy.
* Presence of evaluable disease
* Adequate bone marrow and organ function:

  * Absolute neutrophil count (ANC) ≥1,000 cells/mcL, unless felt to be secondary to underlying MCL (minimum ANC 500 cells/mcL)
  * Hgb ≥ 8 g/dL without transfusional support for 7 days before first treatment, unless felt to be secondary to underlying MCL (minimum Hgb 7.0 g/dL) without transfusional support for 7 days before first treatment)
  * Platelet count ≥50,000 cells/mcL without transfusional support for 7 days before first treatment, unless felt to be secondary to underlying MCL (minimum platelet count 25,000 cells/mcL) without transfusional support for 7 days before first treatment)
  * Renal function assessed by calculated Cockcroft-Gault creatinine clearance (CrCl; see Appendix A) ≥ 30 ml/min. See lenalidomide Treatment Plan, (Table 10-1), for lenalidomide dose adjustment for CrCl ≥ 30 mL/min and < 60 mL/min
  * Adequate hepatic function as determined by:
* Total bilirubin ≤1.5X upper limit of normal (ULN) unless secondary to Gilbert's syndrome or documented liver involvement by lymphoma. Patients with Gilbert's syndrome or documented liver involvement by lymphoma may be included if their total bilirubin is ≤ 5 x ULN
* Aspartate aminotransferase (AST, SGOT) and alanine aminotransferase (ALT, SGPT) ≤ 3 x ULN or ≤ 5 x ULN in cases of documented liver involvement.
* Willingness to receive adequate prophylaxis and/or therapy for thromboembolic events, unless contraindicated in the opinion of the investigator.
* Willingness to undergo confirmatory procedures for assessment of disease status and experimental studies as required by protocol, including bone marrow (BM) aspiration/biopsy and gastrointestinal endoscopy/colonoscopy with biopsy, and/or biopsy of other tissue when appropriate and medically feasible.
* Each patient must sign an informed consent form indicating that he or she understands the purpose of and procedures required for the study and are willing to participate.Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be eligible.
* Willingness of patients who can become pregnant, according to Revlimid/lenalidomide Risk Evaluation and Mitigation Strategy (REMS) criteria, to undergo pregnancy testing in accordance with REMS requirements
* Willingness of all patients to complete surveys and adhere to contraception requirements mandated by the Revlimid/lenalidomide REMS
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate methods of contraception, including at least one method with a failure rate of <1% per year, for at least 28 days prior to Day 1 of Cycle 1, during the treatment period (including periods of treatment interruption), and for at least 2 months after the final dose of glofitamab, 28 days after the last dose of lenalidomide, 18 months after the last dose of obinutuzumab.
* For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 2 months after the final dose of glofitamab, 28 days after last dose of lenalidomide, 6 months after the last dose of obinutuzumab. Men must refrain from donating sperm during this same period.
* Life expectancy ≥ 12 weeks as determined by patient's primary clinician

Exclusion Criteria:

* Investigational agent or anticancer therapy within 5 half-lives prior to start of study therapy except therapeutic monoclonal antibody treatment must be discontinued a minimum of 4 weeks prior to study therapy. An exception is BTKi therapy, which can be continued to prevent disease flare up until 1 day prior to start of study therapy.
* Major surgery within 4 weeks prior to planned start of study therapy.
* Radiotherapy within 7 days of the start of study therapy.
* CART infusion within 30 days prior to Day 1 of Cycle 1
* Active hepatitis B or C, as defined below:

  * HBV surface antigen positive
  * HBV surface antigen negative, HBV core antibody positive and detectable HBV viral DNA. Note: subjects who are HBV core antibody positive and viral DNA negative are eligible. (Prophylactic anti-viral treatment is required for subjects who are HBV core antibody positive)
  * HCV antibody positive and HCV RNA positive.
* History of human immunodeficiency virus (HIV) unless all of the following criteria are met:

  * CD4+ T cell count ≥ 250 cells/mcL
  * No acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within 1 year prior to signing Informed Consent Form
  * Stable (no change in regimen for ≥ 4 weeks) and effective antiretroviral regimen, and HIV viral load < 400 copies/mL within 4 weeks prior to signing Informed Consent form
* Active concurrent malignancy requiring active therapy within the last 3 years with the exception of basal cell carcinoma limited to the skin, squamous cell carcinoma limited to the skin, carcinoma in situ of the cervix or breast, adequately treated lentigo maligna melanoma, or localized prostate cancer. Adjuvant or maintenance therapy to reduce the risk of recurrence of other malignancy previously treated for curative intent is permitted.
* Pregnant or lactating, intending to become pregnant, or unable/unwilling to comply with pregnancy testing and birth control measures and REMS enrollment, as described in inclusion criteria.
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to cycle 1, day 1.
* Clinically significant history of liver disease, including active viral or other hepatitis or current uncontrolled alcohol use disorder that would compromise patient's ability to safely participate in the trial, per clinician's judgment
* Active central nervous system (CNS) involvement with lymphoma, either parenchymal or leptomeningeal
* Presence of ≥Grade 2 toxicity (CTCAE v5.0) due to prior cancer therapy
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Patient with history of confirmed progressive multifocal leukoencephalopathy (PML)
* History of hypersensitivity to compounds of similar biological or chemical composition to IMiDs® and/or the excipients contained in the study drug formulations
* Previous treatment with bispecific antibody therapy directed against CD20 and CD3
* Previous treatment with lenalidomide or other IMiDs® within 12 months of treatment initiation on this study.
* Documented refractoriness to lenalidomide, defined as no response (PR or CR) within 6 months of therapy
* Autologous stem cell transplantation (ASCT) within the period ≤3 months prior to the signing of the informed consent form. Patients with a more distant history of ASCT must exhibit full hematologic recovery before enrollment into the study
* Allogenic stem cell transplantation within the period of ≤3 months prior to signing of the Informed Consent form, evidence of graft-versus-host-disease (GVHD), or receiving active immunosuppression for GVHD.
* A history of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia or are at a high risk for a thromboembolic event in the opinion of the investigator and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period
* Concurrently use other anticancer or experimental treatments
* Administration of a live vaccine within 28 days prior to the start of study treatment (Cycle 1 Day 1).
* Prior treatment with systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents), within 2 weeks or five half-lives (whichever is shorter) prior to first dose of study treatment
* Corticosteroid therapy within 2 weeks prior to first dose of study treatment, with the following exceptions:

  * Short course systemic corticosteroids (total daily dose equivalent of prednisone 100mg or dexamethasone 20 mg) is permissible for disease control, improvement of performance status, or non-cancer indication if administered for ≤ 5 days, and must be discontinued prior to study initiation of study treatment. When clinically indicatedfeasible, tumor assessments such as imaging and biopsies should be performed prior to steroid administration, though this is not required for enrollment.
  * Chronic corticosteroid use of ≤20 mg prednisone equivalent per day, on a stable dose for ≥4 weeks prior to registration.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety, or affect compliance with the protocol or interpretation of results.
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV or Objective Assessment Class C or D cardiac disease, myocardial infarction ≤ 6 months from registration, symptomatic congestive heart failure, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
* Known or suspected chronic active Epstein-Barr viral (CAEBV) infection or reactivation of a latent infection prior to enrollment. CAEBV is a progressive disease with markedly elevated levels of EBV DNA in the blood and infiltration of organs by EBV-positive lymphocytes along with fever, lymphadenopathy, splenomegaly, EBV hepatitis and/or pancytopenia.

  * Participants with detectable EBV titers (quantified using Real-Time qPCR) that are below the level of quantification are eligible.
  * Participants with an EBV titer of <500 IU/mL are eligible, provided that levels are measured monthly for the first 3 months. If there is a rise in EBV levels >500 IU/mL during treatment, management and any therapy should follow local guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2028-01-08 (Estimated); Study Completion 2028-01-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who successfully receive glofitamab | 1 year
  Treatment feasibility defined as the proportion of participants who successfully receive glofitamab during cycles 1-3 without any dose delays of glofitamab for greater than 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kumar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - Dana Farber Cancer Institute (Data Collection and Specimen Analysis), Boston, Massachusetts
  - Mayo Clinic (Data Collection Only), Rochester, Minnesota
  - Washington University (Data Collection Only), St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org